CLINICAL TRIAL: NCT06351202
Title: Impact Assessment of Abdominal Massage on the Feeding Tolerance of Preterms (Less Than 34 Weeks of Amenorrhea) : a Randomized, Single-blind Controlled Trial
Brief Title: Impact Assessment of Abdominal Massage on Feeding Tolerance of Preterms
Acronym: PREMABDO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RBGP 2023 COLNE; 2023-A02256-39 (Other: ANSM)
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2024-05-22 (Actual); Status verified 2024-01

CONDITIONS: Preterm Birth Complication; Digestive System Disease
Keywords: physiotherapy; abdominal massage
MeSH Terms: conditions — Digestive System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- No abdominal massage group (No Intervention): During 14 days, preterm infants with feeding intolerance will not be massed by physiotherapists.
- Abdominal massage group (Experimental): At least 10 abdominal massages will be performed on preterms, by a physiotherapist trained in this technique over a period of 14 days, at the rate of one massage per day.
  Interventions: Other: Abdominal massage

INTERVENTIONS:
Other: Abdominal massage — An abdominal massage for premature babies lasts 10 minutes. Our abdominal massage techniques is described in our protocole and will be adapted according to the term of the child.
  Arms: Abdominal massage group

SUMMARY:
Every year in France, 60,000 children are born prematurely (before 37 weeks of amenorrhea - WA), and present an immaturity of their various systems, in particular the digestive system. This can result in feeding intolerance, expressed by abdominal distension, regurgitation, irregular transit and abdominal discomfort. It can influence the length of hospitalization and lead to necrotising enterocolitis, a major complication.

At the Clermont-Ferrand University Hospital Center, abdominal massages have been performed by physiotherapist for several years in order to improve the state of the digestive system of preterm infants. The indication for abdominal massages are very dependent on the caregivers in charge of the newborns because the evaluation of feeding intolerance remains subjective.

In this context, the investigators carried out a first study to validate a scale that they created (ECAP scale : Clinical Assessment Scale for Abdominal state of Preterm infant) to assess in a rapid, reliable and reproductible manner the abdominal state of preterm infant - data currently being published). This scale can pose the indications for abdominal massage more objectively.

The hypothesis is that abdominal massage improves feeding tolerance (decrease ECAP score), allows faster weight gain and reaching the full ration and therefore reduces the length of hospitalization of preterm infants.

The aim of the study is to assess the effectiveness of abdominal massage, over a period of 14 days, on the feeding tolerance of preterm infants (under 34 weeks of amenorrhea), defined by the achievement and maintenance of an ECAP score less than 4 during 3 days.

DETAILED DESCRIPTION:
This is a single-blind, randomized controlled study. The children will be recruited in the Neonatal Intensive Care Units of the investigation center, by the nursing staff carrying out the ECAP assessment (physiotherapists, nurses, doctors).

An information note will be presented and explained by an element of the medical or paramedical staff to the parents. After a 24 hours reflexion period and answer to any questions they may have, written and informed consent will be requested from both parents for their child's participation in this study.

After obtaining the signed consents, the randomization will follow. In the first group, preterm infants with feeding intolerance will not be massed.

In the second group, at least 10 abdominal massages will be performed by a physiotherapist trained in this technique over a period of 14 days, at the rate of one massage per day.

Each day, the ECAP assessment will be performed at t0min (just before performing an abdominal massage in the massed group) and at t10min (just after performing the massage). The investigators estimate that an abdominal massage for premature babies lasts 10 minutes. The abdominal massage techniques will be adapted according to the term of the child.

ELIGIBILITY:
Inclusion Criteria:

* Newborn, premature, less than 34 Weeks of Amennorhea
* at least 3 days of life
* hospitalized in neonatal intensive care units
* with feeding intolerance demonstrated by an ECAP (Clinical Abdominal Assessement scale for preterms) score equal to or greater than 4/20
* whose holders of parental authority are able to give free and informed consent to participate in this study.

Exclusion Criteria:

* premature newborns with a congenital pathology such as malformation, genetic or chromosomal abnormality
* newborns whose holders of parental authority are protected by law (under guardianship, curatorship, placed under judicial safeguard) or aged under 18
* rejection of participation by parents
* newborns with a contraindication to abdominal massage (fever, major hemodynamic instability)

Ages: 3 Days to 60 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2024-05-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Clinical Abdominal assessment scale for Preterm infants score (ECAP score) | twice day during 14 days
  score between 0 and 20

SECONDARY OUTCOMES:
Variation of the ECAP score (Clinical Abdominal assessement scale for preterms score) between t0 minute and t10 minutes | up to 14 days
  score between 0 and 20
Weight gain of preterm infants with feeding intolerance | up to 28 days
  Daily weight of preterm infants, in z-score
Duration to reach the full ration | up to 28 days
  Number of days needed to reach the full ration (120mL/kg/day)
Duration of hospitalization in level 3 | up to 3 months
  Total number of days of hospitalization in level 3
6-hour fasting windows | up to 28 days
  Number of 6-hour fasting windows
Incidence of occurrence of necrotizing enterocolitis | up to 28 days
  number of necrotizing enterocolitis
Evolution of digestive tolerance over time | up to 28 days
  Raw ECAP value at t10 minutes over time

CONTACTS AND LOCATIONS:
Locations (1):
- CHU clermont-ferrand, Clermont-Ferrand, France